CLINICAL TRIAL: NCT04025346
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Efficacy of Capsimax on Metabolic Rate
Brief Title: To Evaluate the Efficacy of Capsimax on Metabolic Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: OM/190402/CAPSIMAX
Record Dates: First submitted 2019-07-08; First posted 2019-07-18 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2019-12

CONDITIONS: Metabolism

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsimax (Active Comparator)
  Interventions: Other: Capsimax; Other: Micro Crystalline Cellulose
- Placebo (Placebo Comparator)
  Interventions: Other: Capsimax; Other: Micro Crystalline Cellulose

INTERVENTIONS:
Other: Capsimax — 1 capsule to be taken before breakfast.
Other: Micro Crystalline Cellulose — 1 capsule to be taken before breakfast.

SUMMARY:
Capsimax™ is a proprietary Capsicum Extract that employs Beadlet Technology. In the previous study it has been used to investigate its effect in reducing body fat/weight and increase metabolic rate. In this study, Capsimax™ will be used to assess effect on Resting Energy Expenditure (REE) using Indirect Calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male/female participants with age ≥ 18 ≤ 55 years.
* A Body Mass Index (BMI) between 18.5 to 29.9 kg/m2.
* Fasting blood sugar ≤ 100 mg/dl
* Hemoglobin: Males ≥ 11 g/dl and Females ≥ 10 g/dl
* BP < 140/90 mmHg

Exclusion Criteria:

* Post-menopausal females
* History of hypo/ hyperthyroidism.
* History of significant neurological or psychiatric condition such as seizures, depression, or insomnia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Effect of Investigational Product on Resting Energy Expenditure | From baseline to 4 hours.
  Assessed by Indirect Calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Vedic Lifesciences Pvt. Ltd., Thane, Maharashtra, India